CLINICAL TRIAL: NCT05926830
Title: Extracorporeal Flow Abolition in Relation With Primary Insufficiency of Great Saphenous Veins (GSV) Using High Intensity Focused Ultrasound (HIFU) Generated by Sonovein: A Multi Center Prospective Pivotal Study (VEINRESET)
Brief Title: Extracorporeal Flow Abolition in Relation With Primary Insufficiency of Great Saphenous Veins (GSV) Using High Intensity Focused Ultrasound (HIFU) Generated by Sonovein: A Multi Center Prospective Pivotal Study
Acronym: VEINRESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-VN-FDA-VEINRESET 01
Record Dates: First submitted 2023-06-14; First posted 2023-07-03 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Chronic Venous Insufficiency
Keywords: Varicose Vein; HIFU; Theraclion
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sonovein Treatment (Experimental)
  Interventions: Device: Sonovein Treatment

INTERVENTIONS:
Device: Sonovein Treatment — The Sonovein System provides High Intensity Focused Ultrasound (HIFU) ablation of soft tissue. The energy is delivered via an extra-corporeal treatment probe, which includes an imaging system. The high-energy ultrasound waves propagate through the skin and are focused on a portion of the target tissue, generating intense heat and causing local cell apoptosis and progressive tissue volume reduction over the following months in the tissue. The process is then repeated in a stepwise fashion.

SUMMARY:
This is a multi-center series assessment with a planned accrual of 70 patients with diagnosed symptomatic primary GSV insufficiency. Patients will be consented at a Pre-Study Visit and evaluated for eligibility and for baseline characteristics of the disease. Patients will receive treatment with Sonovein for the targeted segments of GSV. At follow-up visits at 7 days (1 to 10 days), 3 months (+/- 20 days), 6 months (+/- 25 days), and 12 months (+/- 30 days) changes in veins and flow characteristics will be evaluated by ultrasound, and patient well-being, including pain which will be evaluated by patient-reported VAS evaluations. Continued follow-up for a total of 12 months will be completed prior to subject study exit. Adverse events (AE) will be assessed at every study visit following HIFU treatment.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for venous procedure with primary GSV insufficiency involving reflux in the segment to be treated
* CEAP-clinical classification ≥ 2
* Physical condition allowing ambulation after the procedure.
* Agree to comply with the Clinical investigation plan and follow-up schedule of the study
* Targeted tissue reachable for treatment with the device.
* Age over 22 years at the time of enrollment.
* No acute venous thrombosis.
* No complete or near complete deep vein post-thrombotic disease.
* Patient has signed and understood the written informed consent.

Exclusion Criteria:

* Patient is pregnant
* Known allergic reaction to anesthetics to be used.
* Legally incapacitated or imprisoned patients
* Patient's vein target not clearly visible on the ultrasound images (in B mode) at the inclusion visit
* Patient participating in another clinical trial involving an investigational drug or device.
* Ankle-brachial index <7 (ABI)
* Undergoing active anticoagulant therapy within the last 6 months
* Diameter of the treated anatomical segment below ≤ 2mm & above > 20mm
* Patients where HIFU cannot be delivered to tissues where macro calcifications induce a significant shadow in the ultrasonic image
* Patients where EPack must be put in contact with an ulcer
* Patients with significant thick scars on the skin over the segment to be treated
* Security distance respected in regards of :

  * nerves & bones
  * the surrounding vessels
* Patient who may not be considered as good candidates for treatment by the investigator outside the explicit exclusion criteria above listed

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Vein Occlusion Rate | 12 months
  Percentage of limbs with occlusion of the treated vein (as measured by Duplex ultrasound)

SECONDARY OUTCOMES:
Complications | 12 months
  Number of limbs presenting complications and side effects resulting from the GSV intervention
Reflux-free Rate | 12 months
  Percentage of limbs without reflux in the treated vein (as measured by Duplex ultrasound)
Venous Clinical Severity Score (VCSS) | 12 months
  Assessment of venous disease (Scale 0-30: MIN=0 (least severe); MAX=30 (most severe))
Clinical-Etiology-Anatomy-Pathophysiology (CEAP) | 12 months
  Clinical signs and symptoms of lower limb venous disease (Scale C0-C6: MIN: C0=no visible or palpable signs of venous disease; MAX: C6=active venous ulcer)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Englewood Health, Englewood, New Jersey
  - Northwell Health, Lake Success, New York
- Praxis für Phlebologie, Melk, Austria
- Phlebomedica s.r.o, Říčany, Czechia

IPD SHARING:
Plan to Share IPD: No